CLINICAL TRIAL: NCT02384213
Title: Incidence of and Prognostic Factors Associated With Heart Failure Following Myocardial Infarction (iHF): a CALIBER Study
Brief Title: Incidence of and Prognostic Factors Associated With Heart Failure Following Myocardial Infarction: a CALIBER Study
Acronym: iHF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: 14_198R
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure; Myocardial Infarction
MeSH Terms: conditions — Heart Failure; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objectives of this study are: i) to investigate the incidence and prevalence of fatal and non-fatal heart failure (HF) following myocardial infarction (MI) and its evolution over time in men and in women; ii) to identify prognostic factors for developing HF in patients who had an MI.

DETAILED DESCRIPTION:
Heart failure (HF) is a major medical problem in the western world. Heart failure is associated with a substantial morbidity and mortality and contributes to a significant extent to economic loss for healthcare systems. An increased prevalence of HF is expected as survival is increasing after an ischaemic event due to primary percutaneous coronary intervention (PCI) and due to demographic changes (ageing population). At this moment, no contemporary data of large scale electronic health records cohorts have been reported regarding the incidence of HF following myocardial infarction (MI). The aim of this research is to investigate the incidence of HF following MI across different time periods and search for predictors of HF following MI to identify high-risk patients. Using CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) data, patients with HF following MI will be identified and the incidence of HF after MI will be described. Prognostic factors associated with the occurrence of HF in patients having experienced a MI will be studied. This is important for future observational research, clinical trials, measuring health outcomes and guideline development.

The study has two aims. First to describe the 'real-world' incidence of HF following MI. Differences between clinically relevant groups (e.g. men and women, and patients with or without - ST-elevation MI,) will be examined. Second, to identify prognostic factors for developing HF in patients who had an MI. The following panels of prognostic factors will be investigated: sociodemographic; anthropomorphic and haemodynamic; behavioural; co-existing conditions (cardiovascular and non-cardiovascular); blood biomarkers; prescribed secondary preventive medication.

This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the NIHR and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (CPRD) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a coded diagnosis for myocardial infarction in their primary or secondary care record.
* Patients in CPRD practices which are deemed "up to standard" for more than 1 year by CPRD criteria.
* Patients with at least one year of follow-up in the CPRD practice CPRD.

Exclusion Criteria:

* A past medical history of heart failure before index MI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adults aged 18 years and over, registered in CPRD practices in England consenting to data linkage, with at least one year of validated pre-study follow-up data, and who experienced a first MI recorded in CALIBER from 1998 to 2010 are potentially eligible.
  Definition MI: MI as recorded in HES or ONS (ICD-10 codes I21-I23), CPRD or MINAP. The type of MI (ST-elevation MI, STEMI; non ST-elevation MI, NSTEMI; or MI not otherwise specified) is coded in MINAP and CPRD.
  Patients will be right censored at end-of-study, which corresponds to the administrative censoring date of the CPRD dataset, patient death or patient deregistration from the general practice.
Sampling Method: Non-Probability Sample
Enrollment: 55000 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Heart failure | Throughout follow-up (maximum 12 years)

SECONDARY OUTCOMES:
Non-cardiovascular mortality | Throughout follow-up (maximum 12 years)
Cardiovascular mortality | Throughout follow-up (maximum 12 years)
Myocardial infarction | Throughout follow-up (maximum 12 years)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Hemingway, FRCP, Study Director — University College, London; Folkert W. Asselbergs, MD, PhD, Principal Investigator — University College, London
Locations (1):
- Farr Institute, University College London, London, United Kingdom